CLINICAL TRIAL: NCT06480188
Title: Differences in Brain Network Mechanisms Between STN and GPi Deep Brain Stimulation
Brief Title: Differences in Brain Network Mechanisms Between STN and GPi Deep Brain Stimulation in the Treatment of Craniocervical Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024KY-102
Record Dates: First submitted 2024-06-14; First posted 2024-06-28 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Device: Deep Brain Stimulation (DBS) of Gpi，PINS G106R Device: Deep Brain Stimulation (DBS) of STN，PINS G106R
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): GPi-DBS group
  Interventions: Device: deep brain stimulation
- Group B (Experimental): STN-DBS group
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation — Group A was the GPi-DBS stimulation group； Group B was the STN-DBS stimulation group

SUMMARY:
Craniocervical dystonia, characterized by symptoms distributed in the craniofacial and/or cervical regions, is a type of focal or segmental dystonia and is the most common form of dystonia in adults. Deep brain stimulation (DBS) is a significant therapeutic approach for medically refractory craniocervical dystonia. The commonly utilized DBS targets are the Globus Pallidus internus (GPi) and the Subthalamic Nucleus (STN). Current research indicates no significant difference in efficacy between these two targets, although there are some differences in the onset time, stimulation voltage, and complications. Studies utilizing magnetic resonance imaging (MRI) to assess brain activity differences in patients with dystonia have found that patients exhibit increased activity and enhanced plasticity across a broad range of brain regions, including the brainstem, cortex, subcortical structures, and the basal ganglia, among others. Consequently, an increasing number of studies are classifying dystonia within the spectrum of brain network disorders. This study aims to recruit patients with craniocervical dystonia who meet the inclusion criteria, randomly assigning them into two groups of 30 patients each. One group will receive stimulation targeting the STN, and the other will target the GPi. Using functional MRI, researcher will conduct a dynamic brain network analysis to explore the differences in the brain network mechanisms underlying the treatment of craniocervical dystonia patients between the STN and GPi targets.

DETAILED DESCRIPTION:
The objectives of this study are: 1) to explore the differences of brain network mechanisms between STN and GPi targets in craniocervical dystonia; 2. To explore the effects of DBS on dysarthsia and dysphagia in patients with craniocervical dystonia and the differences in efficacy, quality of life and side effects between GPi and STN targets in the treatment of craniocervical dystonia; 3. To explore the differences in the electrophysiological signals of nuclei collected during DBS surgery and their application in programming.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Meeting the diagnostic criteria for primary craniocervical dystonia (including patients with cranial, cervical, or unilateral extremity dystonia)
3. Disease duration ≥1 year
4. Normal cognitive function
5. The subject himself or his legal representative can sign the informed consent form

Exclusion Criteria:

1. Patients with other dystonia who did not meet the inclusion criteria
2. Diagnosed with other neuropsychiatric diseases (Alzheimer's disease, amyotrophic lateral sclerosis, Parkinson's disease, etc.)
3. Previous history of craniocerebral surgery
4. Major depression or anxiety
5. The presence of neurosurgical contraindications such as cerebral infarction, hydrocephalus, cerebral atrophy, and sequelae of cerebrovascular disease
6. Contraindications to CT/MRI scanning (e.g. Claustrophobia)
7. women known to be pregnant or lactating, or who had a positive pregnancy test before randomization
8. Presence of contraindications to general anesthesia (such as severe arrhythmia, severe anemia, abnormal liver and kidney function, etc.)
9. Expected survival less than 12 months
10. has participated in other interventional clinical studies that may have affected the outcome assessment
11. other circumstances considered by the investigator to be inappropriate for participation in the study or likely to pose a significant risk to the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
resting-state functional magnetic resonance imaging data | Change from baseline at 1, 6，12 months and 24 months
  First, all participants underwent a standardized rs-fMRI scan for data collection of resting-state BOLD signals. Secondly, data preprocessing was carried out, including head movement correction, non-brain tissue removal, temporal layer correction, spatial normalization, filtering, and removal of physiological noise. Then, the brain network was constructed based on the pre-processed data and the structural features of the brain network were identified. Finally, statistical analysis was used to compare the differences in brain network characteristics between the two groups.

SECONDARY OUTCOMES:
Burke-Fahn-Marsden Scale (BFMDRS) | Change from baseline at 1, 6，12 months and 24 months
  This scale was used to evaluate the severity of dystonia in the subjects, with a total score of 120 points, with higher scores indicating greater symptom severity
Toronto West Spasmodic Torticollis Rating Scale Scale(TWSTRS) | Change from baseline at 1, 6，12 months and 24 months
  The total score ranges from 0 to 85, with higher scores indicating more severe disease symptoms
Craniocervical Dystonia Questionnaire | Change from baseline at 1, 6，12 months and 24 months
  The questionnaire each entry into 0 (never) - 4 points (always), higher scores on behalf of the increasingly serious damage
Frenchay dysarthria scale | Change from baseline at 1, 6，12 months and 24 months
  The scale is divided into 28, each fine items according to the severity was divided into a to e grade 5
Watian Drinking Experiment | Change from baseline at 1, 6，12 months and 24 months
  The Watian Drinking Experiment was used to evaluate the swallowing function of the subjects on a 5-point scale, and the normal level was 1 (swallow water within 5 seconds). Suspicious for level 1 (more than 5 seconds will swallow water) or level 2; Exception for 3 ~ 5
Number of Deep Brain Stimulation programming | Change from baseline at 1, 6，12 months and 24 months
  The number of times participants were programmed after DBS
Number of side effects in Deep Brain Stimulation programming | Change from baseline at 1, 6，12 months and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ustc, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No